CLINICAL TRIAL: NCT04812041
Title: Relationship Between Delirium Severity by CAM-ICU 7 and 4C Mortality Score of the COVID-19 Patients in ICU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, ismail aytaç, medical doctor, Ankara City Hospital Bilkent
Other Study IDs: E1-21-1461
Record Dates: First submitted 2021-03-21; First posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Delirium; Covid19; Intensive Care Unit Delirium
MeSH Terms: conditions — Delirium; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intensive care unit delirium: Covid-19 patients in ICU are screened for delirium and rated the severity with CAM-ICU 7 scores.
  Interventions: Other: CAM-ICU 7 score; Other: 4C Mortality Score

INTERVENTIONS:
Other: CAM-ICU 7 score — A 7-point rating scale (0-7) was derived from the CAM-ICU and RASS assessments 0-2: no delirium, 3-5: mild to moderate delirium, and 6-7: severe delirium.
Other: 4C Mortality Score — 4C Mortality Scores of the patients will be calculated, according to age, gender, number of comorbidities, respiratory rate, SpO2, GCS, urea, and CRP parameters

SUMMARY:
Aim: to investigate whether the 4C Mortality score, which measures the severity of COVID-19, and the CAM-ICU 7 score , which measures the severity of delirium, in ICU. To compare two scores in terms of the number of days without intubation and 28 day mortality rates in ICU.

ELIGIBILITY:
Inclusion Criteria:Patients hospitalized in the intensive care unit diagnosed with COVID-19 will include in the study

Exclusion Criteria:there is no exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in the intensive care unit diagnosed with COVID-19 will participate in the study.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-01-21 (Actual); Primary Completion 2021-05-15 (Estimated); Study Completion 2021-05-25 (Estimated)

PRIMARY OUTCOMES:
28 day mortality | 28 days
  28 day mortality

CONTACTS AND LOCATIONS:
Overall Officials: betül aytaç, MD, Study Chair — ankara ch bilkent
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Khan BA, Perkins AJ, Gao S, Hui SL, Campbell NL, Farber MO, Chlan LL, Boustani MA. The Confusion Assessment Method for the ICU-7 Delirium Severity Scale: A Novel Delirium Severity Instrument for Use in the ICU. Crit Care Med. 2017 May;45(5):851-857. doi: 10.1097/CCM.0000000000002368. PMID 28263192
- [Result] Knight SR, Ho A, Pius R, Buchan I, Carson G, Drake TM, Dunning J, Fairfield CJ, Gamble C, Green CA, Gupta R, Halpin S, Hardwick HE, Holden KA, Horby PW, Jackson C, Mclean KA, Merson L, Nguyen-Van-Tam JS, Norman L, Noursadeghi M, Olliaro PL, Pritchard MG, Russell CD, Shaw CA, Sheikh A, Solomon T, Sudlow C, Swann OV, Turtle LC, Openshaw PJ, Baillie JK, Semple MG, Docherty AB, Harrison EM; ISARIC4C investigators. Risk stratification of patients admitted to hospital with covid-19 using the ISARIC WHO Clinical Characterisation Protocol: development and validation of the 4C Mortality Score. BMJ. 2020 Sep 9;370:m3339. doi: 10.1136/bmj.m3339. PMID 32907855